CLINICAL TRIAL: NCT01580943
Title: Efficacy of Two Commercially Available Chlorhexidine Mouthrinses Non-alcohol Base - a Randomized Clinical Trial
Brief Title: Efficacy of Two Commercially Available Chlorhexidine Mouthrinses Non-alcohol Base
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Daniel Sá Alves, Principal Investigator, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMDUP101351003
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Dental Plaque
Keywords: Chlorhexidine; Cetyl pyridinium chloride; Mouth rinse; Antiplaque Efficacy; Self Efficacy; Taste Sweet; Side Effects
MeSH Terms: conditions — Dental Plaque | interventions — Chlorhexidine; Ethanol; Alkalies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antiplaque Efficacy (Active Comparator): This study was designed as a randomized, two group parallel, double-blind, 3-day non-brushing clinical trial. The sample size (50 participants) was determined using similar studies, making it a convenience sample.
  Over a 72-h experimental non-brushing period, subjects abstained from all forms of mechanical oral hygiene and one group (test) used an 0.12% CHX mouthrinse with 0.05% CPC (Perioaid®), twice daily for 30 seconds and the other group (positive control) used a 0.2% CHX mouthrinse alcohol free (Corsodyl® Care), twice daily for 60 seconds.
  Interventions: Drug: Chlorhexidine
- Taste and Side Effects (Active Comparator): All subjects received a questionnaire using a visual analogue scale designed to evaluate their taste to the mouthrinse, which they had used (What is your opinion concerning the taste of the mouth rinse?). Subjects marked a point on a 10 cm long uncalibrated line with the negative extreme response (0) on the left and the positive extreme (10) at the right end. Then, they were also asked about side effects in an open answer ("Did you feel any side effects caused by mouth rinse?", "If so, what are they?").
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Chlorhexidine — Over a 72-h experimental non-brushing period, subjects abstained from all forms of mechanical oral hygiene and one group (test) used an 0.12% CHX mouthrinse with 0.05% CPC (Perioaid®), twice daily for 30 seconds and the other group (positive control) used a 0.2% CHX mouthrinse alcohol free (Corsodyl® Care), twice daily for 60 seconds. These regimens are suggested by the manufacturers in the instructions
  Other Names: 0,12% CHX with 0,05% CPC (Perioaid®); 0,2% CHX non-alcohol base (Corsodyl® Care)
  Arms: Antiplaque Efficacy
Drug: Chlorhexidine — All subjects received a questionnaire using a visual analogue scale designed to evaluate their taste to the mouthrinse, which they had used (What is your opinion concerning the taste of the mouth rinse?). Subjects marked a point on a 10 cm long uncalibrated line with the negative extreme response (0) on the left and the positive extreme (10) at the right end. Then, they were also asked about side effects in an open answer ("Did you feel any side effects caused by mouth rinse?", "If so, what are they?").
  Arms: Taste and Side Effects

SUMMARY:
The purpose of this study was to compare the antiplaque efficacy of a 0,12% chlorhexidine and 0,05% cetyl-pyridinium chloride mouth rinse (Perio-aid®) with a 0,2% chlorhexidine non-alcohol base mouth rinse (Corsodyl Care®).

DETAILED DESCRIPTION:
Dental plaque is a bacterial biofilm adhering to the tooth surfaces and is not the same in the different areas of the tooth: there is the supragingival, the plaque from the gingival margin and subgingival plaque. It is mainly composed of complex bacterial populations organized in a carbohydrate matrix also containing a small number of epithelial cells, leukocytes, macrophages and inorganic components such as calcium and phosphorus. This biofilm develops in virtually all places where there are damp surfaces and teeth are a very stable support for bacterial colonization. Mechanical oral hygiene procedures such as tooth brushing, dental flossing and inter-dental brushing is the most effective method for plaque removal but mouth rinses containing anti-microbials play an important role in maintaining oral health.

Chlorhexidine (CHX) digluconate, a cationic biguanide, is known to be an effective anti-plaque and anti-inflammatory agent and is the gold standard in chemical plaque control. The benefits of CHX are based on the high intra-oral substantivity and its bactericidal and bacteriostatic activities. This ingredient, when delivered orally, is free from systemic toxicity and microbial resistance, and supra-infections do not occur. It has been proven in several "in vitro" and "in vivo" studies, the safety and long-term efficacy of CHX mouth rinses. There have been suggested many indications for the use of this antiseptic and plaque control is one of the most important factors for proper healing after periodontal surgery and implant therapy.

The 0.2% CHX solution became the standard international concentration, due to his development in Europe but similar levels of plaque inhibition can be achieved with larger volumes of lower concentration solutions of CHX.

A lower concentration of CHX (0.12%) has been tested in several studies and has also been shown to confer clinical benefits. More important than the concentration of CHX seems to be the dose which balances efficacy against local side effects and user acceptability. The optimum dose is considered to be about 20 mg twice daily.

Clinically, the 0,12% CHX have been found to be similarly effective as 0.2% if the volume of the rinse was increased from 10 to 15 ml, yielding an 18 mg dose on each occasion but with respect to plaque growth inhibition, there is a small but significant difference in favour of the 0.2% CHX concentration.

CHX mouthrinses can have a variety of side effects and the most common, according to the manufacturers of these products, are loss of taste, tongue burning and irritation of the oral mucosa. Some brands have lowered the concentration of CHX in their mouthrinses and removed the ethanol in order to eliminate side effects such as soreness and to improve acceptability. A study concluded that the perturbation of taste perception after using 0.12% CHX is significantly lower than that after using 0.2% CHX. On the other hand, another studies concluded that there was no significant difference in terms of taste perception.

This study was a double-blinded, randomized two group parallel, to compare the antiplaque efficacy of two mouth rinses, during a 3-day plaque accumulation model, in periodontal healthy patients. After supragingival prophylaxis participants rinsed twice a day over a 72h non-brushing period. Primary outcome variable was plaque index. As secondary outcomes the taste and side effects variables were studied. Mann-Whitney, χ2 and Fisher's Exact tests were used to compare the variables

ELIGIBILITY:
Inclusion Criteria:

* Good general health without a medical history or medication that might interfere with the conduct of the study
* Dentition with at least 24 teeth (minimum of five teeth per quadrant)
* Periodontal health, pockets < 5mm

Exclusion Criteria:

* Pregnant women or in lactation
* Participants with orthodontic or removable dental appliances
* Known allergies to CHX, CPC or to another ingredient of the mouth rinses
* Systemic antibiotic intake in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
antiplaque efficacy | 72 hours
  antiplaque efficacy of two chlorhexidine mouth rinses: 0,12% chlorhexidine with 0,05% cetyl-pyridinium chloride mouth rinse (Perio-aid®) and a 0,2% chlorhexidine alcohol free mouth rinse (Corsodyl Care®) At baseline, all participants received a through supragingival dental prophylaxis to remove all stain, calculus and plaque.
  After 72h all participants were disclosed with a 1% erythrosine solution and the plaque in both groups was recorded at six sites per tooth on a 5-point scale using the Quigley & Hein (1962) plaque index as modified by Turesky et al. (1970).

SECONDARY OUTCOMES:
taste | 72 hours
  All subjects received a questionnaire using a visual analogue scale designed to evaluate their taste to the mouthrinse, which they had used (What is your opinion concerning the taste of the mouth rinse?). Subjects marked a point on a 10 cm long uncalibrated line with the negative extreme response (0) on the left and the positive extreme (10) at the right end.
Side Effects | 72h
  The participants were asked about side effects in an open answer: "Did you feel any side effects caused by mouth rinse?", "If so, what were they?"

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Alves, DDS, Principal Investigator — Faculdade de Medicina Dentária da Universidade do Porto
Locations (1):
- Faculdade de Medicina Dentária da Universidade do Porto, Porto, Porto District, Portugal

REFERENCES:
- See also: Click here for more information about this study: Efficacy of two commercially available chlorhexidine mouthrinses non-alcohol base - a randomized clinical trial — http://www.fmd.up.pt